CLINICAL TRIAL: NCT00364000
Title: Arterial Stiffness and Arterial Calcifications Evolution in ESRD Haemodialysis Patients Treated by Sevelamer or Calcium Acetate
Brief Title: Arterial Stiffness and Calcifications in Haemodialysis Patients on Sevelamer or Calcium Acetate
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Limitted financial resources
Sponsor: Romanian Society of Nephrology (Other)
Responsible Party: Principal Investigator, Liliana Garneata, MD. PHD, Romanian Society of Nephrology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02_2006
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Haemodialyzed Patients; Hyperphosphatemia
Keywords: haemodialysis; hyperphosphatemia; sevelamer; calcium acetate
MeSH Terms: conditions — Hyperphosphatemia | interventions — calcium acetate; Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Active Comparator): Calcium acetate 670 mg tablets
  Interventions: Drug: Calcium acetate
- II (Experimental): label sevelamer (RenagelR) 800 mg tablets
  Interventions: Drug: Calcium acetate; Drug: Sevelamer

INTERVENTIONS:
Drug: Calcium acetate — Calcium acetate in 240 chronic HD patients
Drug: Sevelamer — label sevelamer (RenagelR) 800 mg tablets
  Arms: II

SUMMARY:
End-stage renal disease (ESRD) is a state of increased arterial stiffness of extensive vessel calcifications, compared with the non-renal population. Both arterial stiffness and arterial calcifications are potent predictors of all-cause and cardiovascular mortality in ESRD patients. Several studies have documented the direct relationship between the extent and severity of arterial/coronary calcifications and outcome in dialysis patients. The relationship is strong no matter if arterial calcifications were quantified by electron-beam computed tomography or a radiological calcification score. Calcifications are early and progressive events in these patients. PWV is strongly related to the degree of sonographic determined arterial calcifications and EBCT-derived coronary artery calcium score in chronic kidney disease patients.

Calcium-based phosphate binders are associated with progressive coronary artery and aortic calcification, especially when mineral metabolism is not well controlled.

According to recent studies, sevelamer hydrochloride is a potent non-calcium-containing phosphate binder, well tolerated in ESRD. Compared with calcium-based phosphate binders, sevelamer is less likely to cause hypercalcemia, low levels of PTH, and progressive coronary and aortic calcification in hemodialysis patients. Moreover, sevelamer has a favorable effect on the lipid profile.

Less is known about the relationship between sevelamer treatment and progression of arterial stiffness. To date, there is one single study examining the influence of sevelamer (versus calcium carbonate) on the evolution of arterial stiffness in a very small number (N=15) of haemodialysis patients. These study used the same patients as historical controls, thus being methodologically rather weak. Moreover, the follow-up was quite short - 6 month.

The aim of the trial is to to quantify, in a randomized opened-labeled controlled trial the effect of sevelamer hydrochloride on the evolution of arterial stiffness parameters (pulse wave velocity and the augmentation index) in chronic haemodialysis patients and to correlate these parameters with arterial calcification assessed by a previous described radiological score of arterial calcification and echocardiographic parameters (left ventricular hypertrophy, LV dilatation, systolic and diastolic dysfunction).

DETAILED DESCRIPTION:
End-stage renal disease (ESRD) is a state of increased arterial stiffness of extensive vessel calcifications, compared with the non-renal population. Both arterial stiffness and arterial calcifications are potent predictors of all-cause and cardiovascular mortality in ESRD patients. Underlying mechanisms for increased stiffness in uremia are not well-defined, but may include: chronic fluid overload, arterial calcifications, microinflammation, increased sympathetic hyperactivity, activation of the renin-angiotensin system, increased lipid oxidation, and abnormalities of the nitric oxide system.

Several studies have documented the direct relationship between the extent and severity of arterial/coronary calcifications and outcome in dialysis patients. The relationship is strong no matter if arterial calcifications were quantified by electron-beam computed tomography or a radiological calcification score. Calcifications are early and progressive events in these patients. PWV is strongly related to the degree of sonographic determined arterial calcifications and EBCT-derived coronary artery calcium score in chronic kidney disease patients.

Calcium-based phosphate binders are associated with progressive coronary artery and aortic calcification, especially when mineral metabolism is not well controlled.

Sevelamer hydrochloride is a potent non-calcium-containing phosphate binder, well tolerated in ESRD. Compared with calcium-based phosphate binders, sevelamer is less likely to cause hypercalcemia, low levels of PTH, and progressive coronary and aortic calcification in hemodialysis patients. Moreover, sevelamer has a favorable effect on the lipid profile.

Less is known about the relationship between sevelamer treatment and progression of arterial stiffness. To date, there is one single study examining the influence of sevelamer (versus calcium carbonate) on the evolution of arterial stiffness in 15 HD patients. These study used the same patients as historical controls, thus being methodologically rather weak. Moreover, the follow-up was quite short - 6 month.

The aim of the study is to quantify, in a randomized opened-labeled controlled trial the effect of sevelamer hydrochloride on the evolution of arterial stiffness parameters (pulse wave velocity and the augmentation index) in chronic haemodialysis patients and to correlate these parameters with arterial calcification assessed by a previous described radiological score of arterial calcification and echocardiographic parameters (left ventricular hypertrophy, LV dilatation, systolic and diastolic dysfunction) 240 chronic clinical stable (young-to-medium-aged)haemodialysis patients will be included. Follow-up: 12 month After screening, the patients will enter a washout period for all currently used phosphate binders for 2 weeks. All patients with hyperphosphatemia (>1.8 mmol/l) during the wash-out period eligible for randomization into the treatment phase.

Stratification will consider the Framingham calcification score, age, gender, diabetes, HD vintage The patient will be randomized (computer-generated) in a 1:1 ratio to open label sevelamer (RenagelR) 800 mg tablets or calcium acetate 670 mg tablets. Because of the size, appearance and taste of the tablets, neither the subjects nor the investigators will be blinded.

Adherence to treatment will be assessed by regular bill count. The starting dose of sevelamer and calcium acetate determined by replacing the phosphate binder used by the patient prior to the washout period on a gram to gram basis. The dose of phosphate binder should be titrated to achieve a serum phosphorus level in the target range of 1-1.6 mmol/L and a serum calcium level <2.6 mmol/L. The maximum elemental calcium dose/day in the calcium acetate arm will not exceed 1.5 g.

Serum ionized calcium will be adjusted for the serum albumin concentration using the formula: adjusted Ca = total measured calcium +0.8 x (4.0-albumin g/dL). After 4 weeks, the dose of phosphate binder, vitamin D analogue and the dialysate calcium concentration can be titrated to reach the target range.

Study conduction will be conducted strictly in compliance with the Declaration of Helsinki and Committees on Human Research in the participating centers/Universities The K/DOQI targets for serum phosphate, serum-calcium and PTH are aimed during the study.

Data on intact parathormone, serum-calcium and phosphate, Ca-P product will be collected monthly in the first three month, every 3 month later on.

Vitamin D allowance only if during the study PTH raise > 500 pg/ml; vitamin D not at all if serum calcium >2.6 mmol/L

Analysis will include:

* correlation between PWV, AIx, calcification scores and Ca-P metabolism parameters, lipid parameters etc
* capability of reaching the N/KDOQI guidelines regarding control of secondary hyperparathyroidism - sevelamer hydrochloride versus calcium acetate
* stratification of PWV and AIx dynamics according to different categories The only published reference in the literature is by Takenaka et al (NDT 2005); they showed in a small study that after 6 months of sevelamer treatment PWV decreases from 14.56 m/s to 13.34 m/s i.e. a decrease of approximatively 9% from pre-Sevelamer values. If normalized to BP (PWV divided by corresponding BP level) than PWV/BP decreased from 10.2 m/s/mmHg to 9.3 m/s/mmHg - i.e. again a decrease of approximatively 9% from pre-Sevelamer values.

Of note, in the previous 6 months, while on CaCO3, PWV increased significantly by 30 to 40% from baseline study values (study of Takenaka has a cross-over design: 6-months on CaCO3 followed by 6-months on Sevelamer). Also there is no information provided on AIx. There is no information in the literature on the impact of Sevelamer on EID (GTN)- vascular function or on EDD (flow-dependent hyperemia or beta2 agonist stimulation)-vascular function.

In our experience, the mean PWV is 7.19+/-1.88 m/s, or if corrected for corresponding BP values: PWV/BP = 5.14 +/- 1.3 m/s/mmHg. AIx is typically 27.9±11.9% in HD patients.

If we assume that the Sevelamer group ("treatment group") will have the same 9% decrease in PWV at 6 months, from baseline, the Ca-binder group ("control group") will have no change (i.e. no increase in PWV - "conservative approach", but different from Takenaka's results where an increase in PWV was reported - see above), the standard deviation of the PWV is 1.88 m/s in our experience or 1.3 m/s/mmHg, the ratio of 1 between the control and thre treatment arms, than for a power of 80% and a confidence interval of 95% we need 108 patients in each arm (105 if PWV/BP is used), 216 total. This will also have sufficient power detect a decrease in AIx of only 4.6% or 16.5% from baseline in the treatment arm. This is usually less than that recorded after different acute interventions (GTN, salbutamol, dialysis session) or after transplantation in HD patients.

Compliance is good in our units and transplantation is rare. Therefore we expect only a dropout rate of 10%. Thus the final study population should be 240 patients. 120 patients should receive Sevelamer for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* more than 3 months on haemodialysis
* willingness to participate
* age 18-60 yrs
* pre-dialysis blood pressure 120-160 mmHg in the last month prior to the initiation of study or recent (<1 Mo) addition of a new antihypertensive drug
* iPTH at entry 200-800 pg/mL (as per severe hyperparathyroidism)
* serum calcium at entry 2.2-2.6 mmol/L

Exclusion Criteria:

* haemodynamic instability
* uncontrolled hypertension
* any severe, debilitating disease associated with a reduced survival
* any major cardiovascular event in the last 12 month before study
* cinacalcet therapy before study entrance
* history of parathyroidectomy
* documented history of poor compliance
* serious gastrointestinal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
changes in arterial stiffness parameters | 6 months
changes in calcification score | 6 months

SECONDARY OUTCOMES:
composite of all-cause mortality, cardiovascular mortality and major cardiovascular events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Covic, Prof, Study Director — "CI Parhon" Clinical Hospital, Iasi; Gabriel Mircescu, Prof, Study Director — "Dr Carol Davila" Teaching Hospital of Nephrology, Bucharest, Romania
Locations (2):
- Romania (2):
  - "Dr Carol Davila" Teaching Hospital of Nephrology, Bucharest
  - "CI Parhon" Clinical Hospital, Iași

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086